CLINICAL TRIAL: NCT00999258
Title: Prospective Trial of Conversion From Tacrolimus to Sirolimus in African American Renal Transplant Recipients With Chronic Allograft Nephropathy
Brief Title: Impact of Conversion From Tacrolimus to Sirolimus in African American Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Serban Constantinescu, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468X1-4504
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Glomerular Filtration Rate; Chronic Allograft Nephropathy
Keywords: glomerular filtration rate; chronic allograft nephropathy; Kidney transplantation; African American
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sirolimus (Active Comparator): the subjects will undergo conversion from tacrolimus to sirolimus OR they will continue to receive tacrolimus.
  Interventions: Drug: sirolimus
- tacrolimus (No Intervention)
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — The subjects assigned to the sirolimus conversion group will be initiated on sirolimus 5mg po daily at which time their tacrolimus dose will be decreased by 50%. Sirolimus levels will be checked within a week and adjusted in a linear fashion to achieve a trough goal of 12-15ng/ml in subjects within 1 year post-transplant, and 8-12 ng/ml in subjects more than 1 year post-transplant. Tacrolimus will be continued in these subjects until sirolimus target trough levels are achieved. Thereafter, tacrolimus will be discontinued indefinitely.
  The subjects assigned to the tacrolimus maintenance group (control group) represent our present standard of care.
  Other Names: GFR measurements and allograft biopsies

SUMMARY:
The objective of this study is to examine the effect on allograft function and histology of converting African American renal transplant recipients with chronic allograft nephropathy (CAN) from a tacrolimus-based regimen to a sirolimus-based maintenance immunosuppression regimen.

The investigators hypothesize that the conversion from tacrolimus to sirolimus in African American renal recipients will stabilize or improve renal allograft function, and stabilize the histological progression of CAN. This conversion will have the potential to prolong long-term graft survival in African American renal transplant patients.

GFR measurements, histological parameters on the allograft biopsy, as well as patient and graft survival, incidence of acute rejection, and specific side effects will be monitored and compared between the sirolimus conversion group and the patients who will be maintained on tacrolimus.

DETAILED DESCRIPTION:
All African American renal transplant recipients (>3months and <5 years post-transplant) at our institution that are currently on a tacrolimus based regimen will be screened. Subjects with 10% or more decrease in glomerular filtration rate (GFR) from baseline, estimated by the MDRD formula,65 and who meet all inclusion criteria will be consented to be enrolled in the study. Baseline will be defined as the highest GFR estimated by MDRD formula, within 3 months of transplant.

Subjects who consent to participate in the study will undergo allograft biopsy and GFR measurement by Gd-DTPA, and will be randomly assigned (2:1) to undergo conversion from tacrolimus to sirolimus or to continue to receive tacrolimus.

The subjects assigned to the sirolimus conversion group will be initiated on sirolimus 5mg po daily at which time their tacrolimus dose will be decreased by 50%. Sirolimus levels will be checked within a week and adjusted in a linear fashion to achieve a trough goal of 12-15ng/ml in subjects within 1 year post-transplant, and 8-12 ng/ml in subjects more than 1 year post-transplant. Tacrolimus will be continued in these subjects until sirolimus target trough levels are achieved. Thereafter, tacrolimus will be discontinued indefinitely. Sirolimus trough levels will be monitored in the study as follows: weekly for the first month, monthly from 1 - 6 months, every 3 months from 6 months - 1 year post conversion. Subjects will continue to receive maintenance immunosuppression consisting of mycophenolate mofetil 500mg to 1000 mg po bid as tolerated and corticosteroid taper per protocol (maintenance of 2.5mg - 5mg po daily at 6 months post-transplant and then indefinitely). GFR measurement by DTPA will be repeated at 6 months, and 1 year post conversion. The second allograft biopsy will be performed at 1 year after sirolimus conversion.

The subjects assigned to the tacrolimus maintenance group (control group) represent our present standard of care. The subjects will continue to receive prednisone, and mycophenolate mofetil, similarly to the subjects assigned to the sirolimus conversion group. In the tacrolimus maintenance group, the subjects will be monitored according to our current clinic protocol, monthly between 3 months - 1 year post transplant, every two months in the second year post-transplant and every 3 months after 2 years. The tacrolimus dose will be adjusted to achieve a trough of 5-10ng/ml in subjects randomized to the control group which is standard of care per protocol. GFR measurement by DTPA will be repeated at 6 months, and 1 year post randomization. The second allograft biopsy will be performed at 1 year post randomization.

Patient and graft survival, and the incidence of acute rejection, proteinuria, hyperlipidemia, anemia, leucopenia, thrombocytopenia, and other clinical parameters will be monitored and compared between the sirolimus conversion group and the subjects who will be maintained on tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* African American (self-identified) renal transplant recipients.
* Primary or re-transplant kidney-only recipients.
* Recipients on tacrolimus-based immunosuppression regimen.
* Time interval after transplant: at least 3 months but not greater than 5 years.
* Renal transplant recipients with 10% decrease in GFR from baseline.
* Women of childbearing potential must have a negative pregnancy test upon enrollment, and must consent to receive contraceptive counseling and to use effective contraception while enrolled in the study. Two reliable forms of contraception must be used simultaneously unless abstinence is the chosen method.

Exclusion Criteria:

* GFR <40ml/min.
* Urine protein-to-creatinine ratio >0.5.
* Significant chronic allograft nephropathy grade 3 Banff score.
* Evidence of acute rejection episodes within the past 3 months.
* Evidence of active infection within the past month.
* Any malignancy except treated non-melanoma skin cancer within the past 3 years.
* Leucopenia <2,000/mm3 within the past month.
* Thrombocytopenia <100,000/mm3 within the past month.
* Total cholesterol >300mg/dl, despite adequate treatment.
* Triglycerides >500mg/dl, despite adequate treatment.
* Non-healed post-surgical or non-surgical wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate measured by Gd-DTPA | 6 months, and 1 year

SECONDARY OUTCOMES:
Quantification the histological markers on renal allograft biopsy | 1 year
Patient survival, graft survival, and incidence of acute rejection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Serban Constantinescu, MD, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States